CLINICAL TRIAL: NCT06592430
Title: The Impact of Communication With Healthcare Providers Via WeChat on Survival Outcomes for Lung Cancer Patietns
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: Wechat-Lung Cancer
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Health Personnel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients diagnosed with lung cancer use WeChat to communicate with healthcare providers
  Interventions: Other: Patients diagnosed with lung cancer use WeChat to communicate with healthcare providers
- Patients diagnosed with lung cancer don't use WeChat to communicate with healthcare providers
  Interventions: Other: Patients diagnosed with lung cancer don't use WeChat to communicate with healthcare providers

INTERVENTIONS:
Other: Patients diagnosed with lung cancer use WeChat to communicate with healthcare providers — Patients diagnosed with lung cancer use WeChat to communicate with healthcare providers
  Groups: Patients diagnosed with lung cancer use WeChat to communicate with healthcare providers
Other: Patients diagnosed with lung cancer don't use WeChat to communicate with healthcare providers — Patients diagnosed with lung cancer don't use WeChat to communicate with healthcare providers
  Groups: Patients diagnosed with lung cancer don't use WeChat to communicate with healthcare providers

SUMMARY:
The use of smartphone-based WeChat applications offers significant advantages in cancer patient education, rehabilitation monitoring, and postoperative symptom management. Through the WeChat platform, patients can access health education materials, engage in online consultations, and interact with doctors and other patients at any time. This ongoing education and psychological support help alleviate patient anxiety and improve their quality of life. This study aims to conduct a prospective observational study in our hospital to explore the impact of WeChat communication on the prognosis of patients with different histological types and stages of lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* (1) Lung cancer patients receiving treatment at Shanghai Pulmonary Hospital (2) ECOG performance status of 0-2 (3) No other serious internal medical conditions (such as severe heart failure, hypertensive crisis, diabetic ketoacidosis, severe liver or kidney impairment, etc.) (4) No history of other malignant tumors in the past 5 years, and no detection of other tumor history during follow-up after lung cancer diagnosis (5) Relevant pathological results

Exclusion Criteria:

* (1) Patients refused enrollment in this study; （2）Patients refused follow-up.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagonosed with lung cacner
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 5 years
  It is defined as the time (years) frome enrollment to death of participants due to an cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date.

IPD SHARING:
Plan to Share IPD: No